CLINICAL TRIAL: NCT00725374
Title: A Exploratory, Double-blind, Randomized, Placebo-controlled Trial to Investigate the Tissue Specific Effects of 2.5 mg Tibolone on Breast Cancer in Postmenopausal Women, in Particular on Breast Tissue Proliferation.
Brief Title: A Study to Investigate the Effects of Tibolone (Livial®) on Breast Tissue in Postmenopausal Women With Breast Cancer (Study 32971)(P06469)
Acronym: STEM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P06469; 32971
Record Dates: First submitted 2008-07-28; First posted 2008-07-30 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — tibolone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Active Comparator): Postmenopausal women of any age, requiring surgery for early invasive primary breast cancer, with estrogen receptor-positive tumor(s). Treated with tibolone
  Interventions: Drug: tibolone
- Arm 2 (Placebo Comparator): Postmenopausal women of any age, requiring surgery for early invasive primary breast cancer, with estrogen receptor-positive tumor(s). Treated with placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: tibolone — one tablet of 2.5 mg tibolone, per day, every day, for 14 ± 2 days (until the day before surgery).
  Other Names: Livial®
  Arms: Arm 1
Drug: placebo — Subjects were to take one tablet of tibolone-matched placebo, per day, every day, for 14 ± 2 days (until the day before surgery).
  Arms: Arm 2

SUMMARY:
The primary purpose of this study is to compare changes in the expression of the proliferation marker Ki-67 in malignant breast tissue after treatment with tibolone or placebo in postmenopausal women who need to undergo surgery for primary breast cancer

ELIGIBILITY:
Inclusion Criteria:

* postmenopausal women of any age
* requiring surgery for early invasive primary breast cancer (clinically stage I or II; T1-T3; N0-1; M0), with estrogen receptor-positive tumor(s)
* body mass index between 18 and 2 kg/m2, inclusive
* must be willing to give voluntary written informed consent.

Exclusion Criteria:

* healthy subjects

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2002-12-15 (Actual); Primary Completion 2005-04-15 (Actual); Study Completion 2005-04-15 (Actual)

PRIMARY OUTCOMES:
The primary objective of this trial was to compare changes in the expression of the proliferation marker Ki-67 in malignant breast tissue after treatment with tibolone or placebo. | The primary outcome measure, the proliferation marker Ki-67, was measured at screening (from the screening biopsy) and about 14 days later (from the surgically removed breast tumour tissue)

SECONDARY OUTCOMES:
Apoptosis index; estrogen/progesterone/androgen receptors & isoforms; bcl-2, bax; pS2; SOX4; Apolipoprotein D; Angiogenesis parameters; estrogen levels, tibolone and tibolone metabolites. | Outcome parameters were measured during the trial as samples were received and at the end of the clinical phase.

REFERENCES:
- [Result] Kubista E, Planellas Gomez JV, Dowsett M, Foidart JM, Pohlodek K, Serreyn R, Nechushkin M, Manikhas AG, Semiglazov VF, Hageluken CC, Singer CF. Effect of tibolone on breast cancer cell proliferation in postmenopausal ER+ patients: results from STEM trial. Clin Cancer Res. 2007 Jul 15;13(14):4185-90. doi: 10.1158/1078-0432.CCR-06-2700. PMID 17634547